CLINICAL TRIAL: NCT00796588
Title: The Effect of Remote Ischemic Preconditioning in Patients Undergoing Major Liver Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Royal Free Hampstead NHS Trust (Other)
Responsible Party: Prof Brian R. Davidson, Royal Free Hospital and Medical School
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: RFH:6100
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Ischemia Reperfusion Injury
Keywords: preconditioning; remote
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients undergoing liver surgery without the designated intervention
  Interventions: Other: remote preconditioning
- RIPC (Other): application of pneumatic tourniquet in patients undergoing liver surgery
  Interventions: Other: remote preconditioning

INTERVENTIONS:
Other: remote preconditioning — Three periods of 10 minute occlusion of blood supply to leg using a pneumatic tourniquet
  Other Names: RIPC

SUMMARY:
The project has been designed to determine whether a brief period of leg ischemia will reduce the I/R injury sustained by the liver during liver surgery and liver transplantation. Adult patients (aged above 18) for liver resection (LR group) and for orthotopic liver transplantation (OLT group) will be analysed separately. Patients from each category will be randomised to two groups - a control and a Remote IPC group. In the remote IPC group Ischemic preconditioning will be induced during surgery by applying a pneumatic tourniquet to the upper part of the right thigh and then inflating it to twice the measured systolic arterial pressure in order to occlude the blood supply of the leg for 10 minutes. The tourniquet will then be deflated for 10 minutes to reperfuse the leg. This is repeated thrice to precondition the skeletal muscles of the leg.

DETAILED DESCRIPTION:
Data Collection & Measurements:

Blood Measurements: Blood will be collected at seven different time points, Baseline, Post IPC, 15 and 90 minutes post IRI and then 6,12 and 24 hours post IRI. At each time point approximately 35 ml of blood will be collected. Samples will be collected for the following measurements: Serum LFT and electrolytes, Serum CPK isozymes, Plasma cytokines, coagulation profile, TEG profile, Plasma cytokines, xanthine and XO/XDH activities, Plasma neutrophil activation, Total plasma Nitrate levels, Plasma lactate and ammonia levels and pulmonary artery blood (from indwelling Swan Ganz) for Plasma Myeloperoxidase levels. Some of these are routine measurements done during and after liver surgery.

Biopsies: Two Liver trucut biopsies - one prior to implantation (and in case of liver resection from the normal remnant liver before occlusion) and the other immediately prior to closure of the abdomen - will be taken to study the changes in tissue oxidation, tissue adhesion molecule upregulation and morphology prior to and after preconditioning.

Intra-operative haemodynamcis: Cardio-pulmonary haemodynamics will be monitored using a Swan-Ganz catheter (if it is clinically indicated and already in place) to note the effects of skeletal muscle ischemic preconditioning on the liver, lungs and the heart. In those patients undergoing liver resection invasive heaemodynamic monitoring will not be performed for the purpose of the study, if not required clinically by the anaesthetists and intensive care physicians. Non-invasive measurements will be made of hepatic and cutaneous circulation using surface Laser Doppler flow meter and Ultra sound probes. Cutaneous microvascular responses to iontophoresis (non-invasive) of acetylcholine, an endothelium-independent vasodilator and sodium nitroprusside, and endothelium-independent vasodilator will be measured using the laser Doppler flow meter. NIRS probes (non -invasive) will be used on the surface of the to measure liver tissue oxygenation. All probes will be properly sterilised prior to application.

Post-operative heamodynamics: Cardio-pulmonary haemodynamics will continue to be monitored using a Swan-Ganz catheter (routinely inserted during liver transplantation) in the post-operative period for 24 hours.

ICG measurements: To assess liver function by injecting 0.5 mg/kg of indocyanine green (ICG) pre-operatively, intra-operatively and post operatively. ICG is routinely used in many liver centres for the assessment of liver function in clinical practise. No additional blood samples will be collected since the uptake and excretion of ICG by the liver will be measured by a non invasive digital pulse densitometric device (ICG Pulsion) connected to the patient by a finger sensor.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 undergoing liver surgery

Exclusion Criteria:

* Absence of written, informed consent.
* Patients with symptomatic peripheral vascular disease and absent or weak peripheral pulses.
* Patients with varicose veins and venous ulcers
* Patients with blood disorders, eg. sickle cell disease
* Patients with any localised limb infections eg. cellulitis
* Pregnancy
* HIV infection
* Fulminant sepsis
* Severe comorbid disease
* Patients below the age of 18

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Does RIPC reduce ischemia reperfusion injury in patients undergoing liver surgery | 8 years

SECONDARY OUTCOMES:
Changes in liver regeneration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Davidson, FRCS, MD, Principal Investigator — Royal Free Hospital and medical School
Locations (1):
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Derived] Robertson FP, Goswami R, Wright GP, Fuller B, Davidson BR. Protocol for a prospective randomized controlled trial of recipient remote ischaemic preconditioning in orthotopic liver transplantation (RIPCOLT trial). Transplant Res. 2016 Apr 6;5:4. doi: 10.1186/s13737-016-0033-4. eCollection 2016. PMID 27054029